CLINICAL TRIAL: NCT04598607
Title: A Multiple-Dose Study to Evaluate the Tolerability and Pharmacokinetics of Hypidone Hydrochloride Tablets in Chinese Healthy Subjects
Brief Title: Tolerability and Pharmacokinetics of Hypidone Hydrochloride in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang Huahai Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HYP104-CTP; 2017ZX09309012 (Other Grant/Funding Number: Ministry of Science and Technology of China)
Record Dates: First submitted 2020-10-13; First posted 2020-10-22 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Hypidone Hydrochloride 60mg (Experimental): 30mg(10mg×3) Hypidone Hydrochloride tablets will be given orally once on day 1, day 9 and twice a day on day 3~8.
  Interventions: Drug: Hypidone Hydrochloride tablets
- Hypidone Hydrochloride 80mg (Experimental): 40mg(10mg×4) Hypidone Hydrochloride tablets will be given orally once on day 1, day 9 and twice a day on day 3~8.
  Interventions: Drug: Hypidone Hydrochloride tablets
- Hypidone Hydrochloride 100mg (Experimental): 50mg(10mg×5) Hypidone Hydrochloride tablets will be given orally once on day 1, day 9 and twice a day on day 3~8.
  Interventions: Drug: Hypidone Hydrochloride tablets
- Placebo 60mg (Placebo Comparator): 3 tablets of placebo will be given orally once on day 1, day 9 and twice a day on day 3~8.
  Interventions: Drug: Placebo
- Placebo 80mg (Placebo Comparator): 4 tablets of placebo will be given orally once on day 1, day 9 and twice a day on day 3~8.
  Interventions: Drug: Placebo
- Placebo 100mg (Placebo Comparator): 5 tablets of placebo will be given orally once on day 1, day 9 and twice a day on day 3~8.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hypidone Hydrochloride tablets — 30mg(10mg×3), 40mg(10mg×4) or 50mg(10mg×5) Hypidone Hydrochloride tablets will be given orally once on day 1, day 9 and twice a day on day 3~8.
  Other Names: HHT101
  Arms: Hypidone Hydrochloride 100mg; Hypidone Hydrochloride 60mg; Hypidone Hydrochloride 80mg
Drug: Placebo — 3, 4 or 5 tablets of placebo will be given orally once on day 1, day 9 and twice a day on day 3~8.
  Arms: Placebo 100mg; Placebo 60mg; Placebo 80mg

SUMMARY:
This study will investigate the tolerability and pharmacokinetics of Hypidone Hydrochloride by multiple doses in 36 healthy male and female subjects who are of 18 to 55 years old.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, randomized, multiple-dose, single center study. 36 male and female healthy subjects will be enrolled in this study. Within 14 days prior to study drug administration, subjects will be screened based on the inclusion and exclusion criteria. The study will be performed in 3 groups of 12 subjects each. In each group of 12 subjects, 10 subjects will be randomly assigned to receive Hypidone Hydrochloride and 2 subjects to receive matching placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese healthy subjects, male to female ratio is 1:1;
2. 18 ≤ age ≤55;
3. Female body weight is not less than 45kg, male body weight is not less than 50kg, BMI is between 18.5~28.0 kg/m2 (including upper and lower limits);
4. Understand and sign informed consent, and participate in clinical trials voluntarily.

Exclusion Criteria:

1. Those who have a history of major diseases such as cardiovascular system, respiratory system, liver, kidney, endocrine system, digestive system, blood and lymphatic system, immune system, nervous system, skeletal system and psychiatry, and who are judged unfit to participate in this study;
2. Any condition or condition that may significantly affect drug absorption, distribution, metabolism, and excretion, such as a history of gastrointestinal surgery (gastrectomy, gastroenterostomy, enterectomy, etc.);
3. General physical examination, vital signs and other abnormalities judged by clinicians as clinically significant;
4. resting pulse rate <55 times/min or >100 times/min;Sitting systolic pressure <90mmHg or >140mmHg, diastolic pressure <60mmHg or >90mmHg;
5. The laboratory examination indicates that the subject has abnormalities that the researcher has determined to be clinically significant;
6. ALT or Cr and BUN exceeding the upper limit of normal value;Urine protein test results "++" or above;
7. Serum virology test (HBs antigen, HCV antibody, syphilis serum reaction (Trust test) and HIV antibody test) with positive results;
8. Abnormal electrocardiogram (ECG) at screening stage is of clinical significance, such as QTc interval ≥450ms in men and QTc interval ≥470ms in women, and the researchers think it is not suitable to be included;
9. patients who had taken any prescription drugs, non-prescription drugs, Chinese herbs, vitamins and other dietary supplements in the two weeks prior to enrollment, and the researchers believe that this situation may affect the evaluation results of this study.
10. Those who have taken food or drink (such as grapefruit) containing enzymes that can induce or inhibit liver metabolism within 1 week before starting the administration of the test;
11. A history of severe allergy or has a history of allergy to two or more foods or drugs;
12. Subjects with a history of smoking 2 weeks before the screening period or subject with positive urine cotinine test during the admission review period;
13. A history of alcohol abuse and consume an average of more than 14 units of alcohol per week (1 unit =285ml beer or 25ml spirits or 150ml wine), or during the study subjects were unable to avoid alcohol consumption within 24 hours before and during the study period or alcohol breath test positive;
14. A history of drug abuse or drug abuse, or those with positive urine drug screening;
15. Pregnant or lactating women;
16. The subject or his/her spouse has a family planning plan within the next 6 months of the last use of the drug, and is unable to use the contraceptive method approved by the Study during the study period as directed by the investigator;
17. Those who had donated blood or lost blood ≥400mL in the 3 months before screening, and those who had donated blood ≥200mL in the 1 month before screening or had a history of component donation;
18. it is impossible to avoid using caffeinated drinks, strenuous exercise, or other factors affecting drug absorption, distribution, metabolism, and excretion within 24 hours before and during the trial;
19. Subjects who have participated in or are participating in other experimental drugs or unlisted drug trials within 3 months prior to screening;
20. Persons directly related to this clinical trial;
21. Subjects who, in the opinion of the investigator, have other factors that are not appropriate to participate in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The ratio of male and female is 1:1.
Enrollment: 36 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Cmax | Day 1-11
  Peak Plasma Concentration
Tmax | Day 1-11
  Time to Peak Plasma Concentration
AUC | Day 1-11
  Area under the plasma concentration versus time curve
T1/2 | Day 1-11
  half-life

SECONDARY OUTCOMES:
Percentage of subjects with treatment-emergent adverse events(TEAE) | Up to Day 15
  Clinical significant Abnormal of Laboratory valuse, physical examination results, vital signs and ECG results will be recorded as TEAE.
Percentage of subjects with abnormal Laboratory values | Up to Day 15
  Laboratory tests including Hematology, Biochemistry and Urinalysis.
Percentage of subjects with abnormal Physical examinations results | Up to Day 15
  Physical examinations including Head and face, skin system, lymph nodes, eyes, ear, nose and throat, mouth, respiratory system, abdomen, cardiovascular system, musculoskeletal and nervous system.
Percentage of subjects with abnormal Vital signs results | Up to Day 15
  Vital signs including sitting blood pressure, pulse rate and ear temperature.
Percentage of subjects with abnormal ECG(12-lead Electrocardiogram) results | Up to Day 15
  ECG tests including heart rates, PR interval, QT interval, corrected QT interval.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China